CLINICAL TRIAL: NCT01201577
Title: Biological Modulation of Bacterial QSSMs, Innate and Adaptive Immunity by Antibiotics, Probiotics and Prebiotics in Healthy Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Dileep Lobob, University of Nottingham
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 09GA014
Record Dates: First submitted 2010-09-13; First posted 2010-09-14 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Quorum Sensing; Prebiotics; Probiotics; Sepsis
Keywords: Quorum sensing; Prebiotics; Probiotics; Sepsis
MeSH Terms: conditions — Sepsis | interventions — Active Hexose Correlated Compound; Azithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo/Probiotic (Active Comparator)
  Interventions: Dietary Supplement: Bifidobacterium longum BB536; Drug: Azithromycin
- Placebo/Prebiotic (Active Comparator)
  Interventions: Dietary Supplement: Active hexose correlated compound (AHCC); Drug: Azithromycin
- Prebiotic/Probiotic (Active Comparator)
  Interventions: Dietary Supplement: Bifidobacterium longum BB536 and Active hexose correlated compound (AHCC); Drug: Azithromycin
- Placebo/Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Corn starch placebo capsule; Drug: Azithromycin

INTERVENTIONS:
Dietary Supplement: Bifidobacterium longum BB536 — 2 capsules od
  Arms: Placebo/Probiotic
Dietary Supplement: Active hexose correlated compound (AHCC) — One capsule tds
  Arms: Placebo/Prebiotic
Dietary Supplement: Bifidobacterium longum BB536 and Active hexose correlated compound (AHCC) — One capsule tds (prebiotic) and two capsules od (probiotic)
  Arms: Prebiotic/Probiotic
Dietary Supplement: Corn starch placebo capsule — One capsule tds and two capsules od
  Arms: Placebo/Placebo
Drug: Azithromycin — 250mg od

SUMMARY:
It has recently been discovered that bacteria are able to communicate using specialised molecules known as Quorum Sensing Signalling Molecules (QSSMs). An accumulation of QSSMs in their surrounding environment allow for the bacteria to quantify the size of colonies. At specific colony sizes the concentration of QSSMs reaches a critical threshold leading to the activation of genes that cause an infection. It is by this mechanism that bacteria within a colony coordinate behaviour to activate infectivity when colony sizes are large enough to withstand defensive measures from the host's immune system. A disruption of quorum sensing may reduce the severity of infection and this has led to the development of inhibitors of quorum sensing as a new strategy in antibacterial therapy.

QSSMs are also thought to facilitate infection by other mechanisms and are able to influence the number and function of a specific type of immune cell known as an 'antigen presenting cell'. These cells are pivotal in allowing the immune system to recognise components of bacteria as foreign and thereby mount the appropriate response. It was found that large numbers of these types of cells underwent programmed cell death (cell suicide) in the presence of QSSMs compared to when QSSMs were absent. This mirrors the situation in blood sampled from patients with severe infections where there is a greater proportion of cell deaths among antigen presenting cells than other types of immune cell.

This study aims to establish in healthy volunteers, the mechanisms by which QSSMs affect immune cells and facilitate the spread of infection. Antibiotic administration in humans can alter the environment of the intestine and can lead to an overgrowth of harmful bacteria to potentially cause an infection. Probiotics supplements can prevent bacterial overgrowth and potentially reduce infective complications. The mechanism, which we aim to clarify, may involve changes in both the production of QSSMs and the function of immune cells.

Hypothesis

1. Antibiotic use alters gut flora, leading to the appearance in the systemic circulation of bacterial QSSMs and changes in immune function of the host.
2. Probiotics and/or prebiotics have beneficial effects by preserving the normal resident gut flora, thereby, modulating bacterial QSSMs and preserving the immune function of the host.

Aims

The aims of our study are 2 fold:

1. Firstly, to study the effect of orally administered antibiotic on QSSMs (in faeces and blood) and on innate and adaptive immunity in healthy humans.
2. Secondly, to study the effect of orally administered combinations of prebiotic, probiotic and antibiotic on QSSMs (in faeces and blood) and on innate and adaptive immunity in healthy humans.

ELIGIBILITY:
Inclusion Criteria:

* Male volunteers
* Age 18-55 years
* Willing to participate and able to give informed consent
* Alcohol abstinence during study

Exclusion Criteria:

* Smokers/substance abusers
* Individuals with diabetes mellitus
* Oral/Intravenous steroids
* Allergy to azithromycin
* Individuals already taking regular medications/probiotics/nutritional supplements
* Individuals with chronic disease or currently under investigation
* Individuals with ≤3 bowel movements/week
* Individuals with ≥2 bowel movements/day

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Serum QSSM level | 14 days

SECONDARY OUTCOMES:
T cell Th1/Th2 ratio | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Abeed Chowdhury, MB ChB BSc MRCS, Principal Investigator — University of Nottingham; Dileep Lobo, MBBS DM FRCS, Study Director — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, Nottinghamshire, United Kingdom